CLINICAL TRIAL: NCT02582723
Title: Acute Effect of Cheeses With Different Energy Content on Appetite
Acronym: STABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Fromageries Bel SA (Industry)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: B323
Record Dates: First submitted 2015-09-17; First posted 2015-10-21 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Appetite; Lack or Loss, Nonorganic Origin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High protein/high fat hard cheese (Active Comparator): Served for breakfast together with bread, juice and coffee, tea or water
  Interventions: Other: High protein/high fat hard cheese
- High protein/low fat hard cheese (Active Comparator): Served for breakfast together with bread, juice and coffee, tea or water
  Interventions: Other: High protein/low fat hard cheese
- Low protein/high fat creme cheese (Experimental): Served for breakfast together with bread, juice and coffee, tea or water
  Interventions: Other: Low protein/high fat creme cheese

INTERVENTIONS:
Other: High protein/high fat hard cheese — Assess whether the cheeses with high protein content have improved effect on satiety compared to the cheese with low protein content.
  Arms: High protein/high fat hard cheese
Other: High protein/low fat hard cheese — Assess whether the cheeses with high protein content have improved effect on satiety compared to the cheese with low protein content.
  Arms: High protein/low fat hard cheese
Other: Low protein/high fat creme cheese — Assess whether the cheeses with high protein content have improved effect on satiety compared to the cheese with low protein content.
  Arms: Low protein/high fat creme cheese

SUMMARY:
A double-blind, randomised crossover design will be employed with three experimental conditions; High protein/high fat hard cheese, high protein/low fat hard cheese, and low protein/high fat creme cheese served at least 7 days apart. After having successfully completed screening procedures, eligible participants will be invited for three separate test days. The test days should be performed at least 7 days apart; however for logistical reasons 4 days can be accepted. On the test days, the products will be provided in a randomized order, and subjective appetite ratings will be measured every 30 minutes for the following 3 hours. Subsequent energy intake will be measured by an ad libitum meal 3 hours following serving of the breakfast meal.

DETAILED DESCRIPTION:
Participants will arrive at the laboratory after an overnight fast (at least from 10:00 pm) with the use of the least strenuously transportation possible (no bicycling or long distance walk). In addition, the preceding two days (48h) before each of the study days; no intensive physical activity or consumption of alcohol is allowed in order to obtain standardization of the participants.

Once settled into an individual feeding cubicle, visual analogue scales (VAS) will be completed for the measurement of fasting appetite levels. A standardized fixed breakfast meal (providing approximately 20% of total estimated energy need) consisting of 80 g. cheese with bread, orange juice and a cup (125 mL) of coffee/the/water (milk is not allowed). The amounts of bread (70.5 g.) and juice (132 g.) are calculated with Babybel original as reference, and these amounts for bread and juice are kept constant regardless of the cheese provided. The cheese will be served blinded together with the bread, and the brand of cheese will not be mentioned for the participants. Participants will be asked to consume this breakfast within 15 minutes and the exact meal duration (in minutes) will be noted after completing the meal in order to examine the eating rate. VAS will be used to measure subjective appetite sensations during the post-meal period as well as the pleasantness of the meal and the study products after completing the meal. VAS will be used to measure subjective appetite sensations for the following hours. Three hours following serving of the breakfast meal, participants will be provided with a homogeneous single item ad libitum lunch meal. The meal is a homogeneous dish of spaghetti bolognese providing a total of 8 MJ and the participants are instructed to eat until they are comfortably full. The energy composition of the meal is 15 E% protein, 30 E% fat and 55 E% carbohydrate. VAS will be used to measure subjective appetite sensations during the post-meal period as well as the pleasantness of the meal after completing the meal. The meal duration (in minutes) will be noted after completing the meal. The ad libitum meal ends the study day, and the participant will be free to leave afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Healthy men and women
* Ages between 18 and 60 years
* BMI between 20.0-31.9 kg/m2
* Regular breakfast eaters (eating breakfast ≥ 4 times a week)
* Regular menstrual periods (women only)

Exclusion Criteria:

* Participants not able to comply with the study protocol, including consumption of the specific study foods
* Significant health problems as judged by the investigator
* Taking any medication or supplements known to affect appetite or body weight within the past month and/or during the study as judged by the investigator
* Pregnant, planning to become pregnant within the next 4 weeks or breastfeeding (women only)
* History of anaphylaxis to food
* Any known food allergies or food intolerance likely to affect the present study
* Smoking, smoking cessation within the past 3 months or nicotine use (electronic cigarettes)
* Self-reporting currently dieting or having lost/gained significant amount of weight (±3 kg) in the previous 3 months
* Significant changes in physical activity patterns in the past 4 weeks or intention to change during the study as judged by the investigator
* Significant change in diet in the past 4 weeks or intention to change the diet during the study as judged by the investigator
* Use of systemic or local treatment likely to interfere with evaluation of the study parameters as judged by the investigator
* Participants who work in appetite or feeding related areas
* Post-menopausal (women only)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Total accumulated energy intake (overall intake of kJ from breakfast and ad libitum meal) | During the three hour study day
  The primary outcome of the study is the total accumulated energy intake including the breakfast meal and the ad libitum test meal.

SECONDARY OUTCOMES:
Feelings of appetite | During the three hour study day
  Secondary outcomes of the study are VAS scores for appetite every 30 minutes throughout the study test days where the feelings of appetite will be analysed in relation to energy content of the meals by calculating satiety quotients.
Pleasantness of meals and test products | After completing each meal at every test day , up to 200 minutes
  Furthermore secondary outcomes are the VAS scores for the pleasantness of the meals after completing each meal as well as the pleasantness of the test products.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Study Chair — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark